CLINICAL TRIAL: NCT00091143
Title: A Pilot Trial of Therapeutic Vaccination With a Modified gp100 Melanoma Peptide (gp100:209-217(210M)), Montanide ISA 51, and KLH With Reconstitution After Chemotherapy to Induce Lymphopenia in Patients With Metastatic Melanoma
Brief Title: Fludarabine Followed by Vaccine Therapy and White Blood Cell Infusions in Treating Patients With Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000383908; PPMC-IRB-02-99; NCI-6361
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2009-08

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; keyhole-limpet hemocyanin; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: keyhole limpet hemocyanin
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Vaccines made from peptides may make the body build an immune response to kill tumor cells. Infusions of a person's white blood cells may be able to replace immune cells that were destroyed by chemotherapy. Combining fludarabine with vaccine therapy and white blood cell infusions may kill more tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects of giving vaccine therapy together with fludarabine and white blood cell infusions and to see how well it works in treating patients with unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity and immune effects of vaccination comprising modified gp100 peptide (gp100:209-217[210M]), Montanide ISA-51, and keyhole limpet hemocyanin followed by peripheral blood mononuclear cell reinfusion after treatment-induced lymphopenia with fludarabine in patients with unresectable or metastatic melanoma.
* Determine the induction of antigen-specific T-cell responses in patients treated with this regimen.
* Determine the kinetics and duration of immune response in patients treated with this regimen.
* Compare the immunologic effects of this regimen in these patients with historical results.

Secondary

* Compare 2 different dosing schedules of fludarabine, in terms of induction of lymphopenia and granulocytopenia and on the induction of a specific immune response to this vaccine, in these patients.

OUTLINE: This is a pilot, randomized study. Patients are randomized to 1 of 2 treatment arms.

Within 2 weeks before the start of fludarabine, all patients undergo leukapheresis over 4-6 hours for the collection of peripheral blood mononuclear cells (PBMCs).

* Arm I: Patients receive fludarabine IV over 30 minutes on days 1-5.
* Arm II: Patients receive fludarabine as in arm I on days 1, 3, and 5. In both arms, patients receive autologous PBMCs IV over approximately 30 minutes on day 8 and vaccination comprising gp100:209-217(210M) peptide, Montanide ISA-51, and keyhole limpet hemocyanin subcutaneously on days 8, 22, 36, 50, and 64. Patients with stable or responding disease continue to receive vaccination on day 78 and then every 28-31 days for up to 1 year.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 20 patients (10 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant melanoma

  * Metastatic or unresectable disease
* Measurable disease
* HLA-A2 positive
* Received at least 1 prior immunotherapy and/or chemotherapy regimen for metastatic disease (first 6 patients only)
* No known brain metastases unless previously treated with radiotherapy and/or surgery AND is stable for at least 1 month after treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Absolute lymphocyte count ≥ 500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusions allowed)
* Hematocrit ≥ 24%
* No other active bleeding

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN) (unless due to Gilbert's disease)
* AST and ALT < 3 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine < 2 mg/dL
* No uncontrolled hypercalcemia

Cardiovascular

* No uncontrolled symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia
* No uncontrolled hypertension

Pulmonary

* No uncontrolled bronchospasm
* No hemoptysis

Immunologic

* Negative serology for all of the following:

  * HIV-1 and HIV-2
  * HTLV-1 and -2
  * Syphilis
* Rheumatoid factor < 43 units/μL
* Anti-nuclear antibody < 11 units/μL
* No history of multiple sclerosis, systemic lupus erythematosus, or myasthenia gravis
* No primary or secondary immunodeficiency
* No active infection
* No allergy to seafood or shellfish that would preclude study participation

Other

* No active gastrointestinal bleeding
* No uncontrolled hyperglycemia
* No other medical or psychiatric condition or social situation that would preclude study compliance
* No other uncontrolled illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3-4 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior immunization with gp100:209-217(210M) peptide

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* More than 2 weeks since prior steroid therapy except replacement steroids or inhaled steroids
* No concurrent corticosteroids except replacement steroids
* No concurrent dexamethasone

Radiotherapy

* See Disease Characteristics
* More than 2 weeks since prior radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Toxicity by clinical and laboratory observation at 1 month
Antigen-specific T-cell responses by tetramer analysis, ELISPOT, and cytokine flow cytometry periodically

SECONDARY OUTCOMES:
Compare 2 different dosing schedules of fludarabine in terms of lymphocyte recovery using a complete blood count periodically
Tumor regression by standard imaging at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Urba, MD, PhD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Research Institute
Locations (1):
- Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon, United States